CLINICAL TRIAL: NCT00893529
Title: A Double-blind, Randomized Trial of the Efficacy of Replacing Sugary Drinks by Low-sugar Alternatives on Body Weight and Fat Mass in School Children
Brief Title: A Study of the Effect of Replacing Sugary Drinks by Low-sugar Alternatives on Body Weight and Fat Mass in Children
Acronym: DRINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Heart Foundation (Other); KNAW: Royal Netherlands Academy of Arts and Sciences (Unknown)
Responsible Party: Principal Investigator, Margreet R. Olthof, Dr ir, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZONMW120520010-NHS2008B096
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Body Weight
Keywords: overweight; children; intervention; sugar-sweetened beverages
MeSH Terms: conditions — Body Weight; Overweight | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dietary intervention 1 (Experimental)
  Interventions: Dietary Supplement: lemonade with sugar
- dietary intervention 2 (Experimental)
  Interventions: Dietary Supplement: lemonade low in sugar

INTERVENTIONS:
Dietary Supplement: lemonade with sugar — 250 milliliters of lemonade with sugar daily for 18 months
  Arms: dietary intervention 1
Dietary Supplement: lemonade low in sugar — 250 milliliters of lemonade low in sugar daily for 18 months
  Arms: dietary intervention 2

SUMMARY:
Obesity results from an imbalance between energy intake and energy expenditure. There is much speculation about foods that are particularly fattening, and sugary drinks are seen as major culprits. It is hypothesized that a high intake of calories from sugary drinks would not be compensated for by reduced food intake at subsequent meals. As a result, body weight would increase. In this double-blind, long term, randomized controlled trial the effect of replacing sugar-containing beverages by low-sugar alternatives on body weight and fat mass in children will be investigated.

DETAILED DESCRIPTION:
Rationale: Liquid carbohydrates (including soft drinks as well as fruit juices) are thought to be less satiating then solid carbohydrates (e.g., bread or fruits). The hypothesis is that calories from sugary drinks might not be compensated for by eating less at subsequent meals and body weight would increase. In this way liquid carbohydrates might be one of the causes of becoming overweight and obesity. However, the evidence for a causal relation between sugary drinks and weight gain is inconclusive.

Objective: To test the effect of replacing sugar-containing beverages by beverages low in sugar on body weight and fat mass in children aged 5-10 years.

Study design: A double-blind, long term, randomized controlled trial.

Study population: Healthy school children in the age of 5-10 years old. We consider it unethical to encourage children to drink sugary drinks. Therefore children are only eligible if they already habitually consume 250 mL per day or more of sugary drinks.

Intervention: Six hundred healthy children (5-10 years) will be divided randomly into 2 groups. Group 1 (n=300) receives 250 mL per day of sugar-containing lemonade. Group 2 (n=300) receives 250 mL per day of lemonade low in sugar. The low-sugar drinks are sweetened with artificial sweeteners. The drinks will be consumed during the morning break during the weekdays at school and at home during weekends and holidays. The intervention period will be 18 months.

Before the main trial starts feasibility and logistics will be tested in a pilot study. The design of the pilot study will be a 2-month randomized controlled trial in approximately 80 school children aged 5-10 years.

Main study parameters/endpoints: The primary outcome of the study is children's body weight (body mass index, corrected for age). Secondary endpoints are waist circumference, skin folds and bioelectrical impedance. These outcomes will be measured four times during the study, at 0, 6, 12 and 18 months. As a secondary outcome we will also perform a sensory evaluation at 0, 6, 12 and 18 months and a questionnaire about dental health at 12 and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy school boys and girls
* Age 5 years and older, children still have to be in elementary school at the end of the study
* Children who already habitually consume 250 mL per day or more of sugary drinks

Exclusion Criteria:

* Using medication or under medical treatment for obesity
* Any acute or chronic disease such as diabetes, growth disorders, celiac disease, or serious gastroenterological diseases
* Medical history or surgical events known to interfere with the study
* Participation in another intervention trial up to 3 months before and during the study, if the intervention interferes with the current study
* Physical disabilities that hamper the measurements
* Intention to change location of residence and primary school during the study period

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 641 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index Z-score | 0, 6, 12, and 18 months

SECONDARY OUTCOMES:
Skinfolds | 0, 6, 12 and 18 months
Waist to height ratio | 0, 6, 12 and 18 months
Bioelectrical Impedance | 0, 6, 12 and 18 months
  % fat mass
Dental health | 12 and 18 months
Sensory evaluation | 0, 6 ,12 and 18 months
  We perform a sensory evaluation, to relate the effects at the end of the trial to properties of our drinks, asking:
  1. How much do you want to drink the study drink?
  2. How satiated do you feel?
  3. What do you eat together with the study drink?
  4. How much do you like the study drink?
  The questionnaire includes pictures, and was tested at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martijn B Katan, Prof. Dr., Principal Investigator — VU University of Amsterdam; Margreet R Olthof, Dr., Principal Investigator — VU University of Amsterdam
Locations (1):
- VU University Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Katan MB, de Ruyter JC, Kuijper LD, Chow CC, Hall KD, Olthof MR. Impact of Masked Replacement of Sugar-Sweetened with Sugar-Free Beverages on Body Weight Increases with Initial BMI: Secondary Analysis of Data from an 18 Month Double-Blind Trial in Children. PLoS One. 2016 Jul 22;11(7):e0159771. doi: 10.1371/journal.pone.0159771. eCollection 2016. PMID 27447721
- [Derived] de Ruyter JC, Katan MB, Kuijper LD, Liem DG, Olthof MR. The effect of sugar-free versus sugar-sweetened beverages on satiety, liking and wanting: an 18 month randomized double-blind trial in children. PLoS One. 2013 Oct 22;8(10):e78039. doi: 10.1371/journal.pone.0078039. eCollection 2013. PMID 24167595
- [Derived] de Ruyter JC, Olthof MR, Seidell JC, Katan MB. A trial of sugar-free or sugar-sweetened beverages and body weight in children. N Engl J Med. 2012 Oct 11;367(15):1397-406. doi: 10.1056/NEJMoa1203034. Epub 2012 Sep 21. PMID 22998340